CLINICAL TRIAL: NCT01635504
Title: Posterior Cheek Enlargement in HIV: Anatomic Characterization and Treatment With Botulinum Toxin A
Brief Title: HIV Posterior Cheek Enlargement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H12-00990
Record Dates: First submitted 2012-06-04; First posted 2012-07-09 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: HIV Posterior Cheek Enlargement
Keywords: HIV lipoatrophy; masseter hypertrophy; parotid enlargement; botulinum toxin
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- botulinum toxin A (Experimental)
  Interventions: Biological: Botulinum toxin A

INTERVENTIONS:
Biological: Botulinum toxin A — Botulinum toxin A 50 units per side of the posterior cheek enlargement, injected into the masseter muscle and parotid gland (10 units into 5 points of the posterior cheek enlargement per side, giving a total of 100 units per patient)
  Other Names: Botox

SUMMARY:
Altered contour of the lower face is a frequent complication of human immunodeficiency virus (HIV). HIV facial lipoatrophy or loss of facial fat commonly results from antiretroviral therapy. Posterior cheek enlargement leading to a bulky and widened lower facial contour can also be seen in HIV. These changes can lead to significant cosmetic disfigurement and have an enormous psychosocial impact on patients. They also make individuals vulnerable by making them recognizable as persons living with HIV. Posterior cheek enlargement has not been well characterized. Both the parotid salivary gland and the masseter muscle are located in the posterior cheek region. Although parotid gland enlargement in a common complication of HIV, it is unknown whether enlargement of the masseter muscle also contributes. The investigators plan to study posterior cheek enlargement in HIV positive individuals. The investigators also plan to use botulinum toxin A as a novel treatment to improve the altered lower facial contour seen in HIV. This treatment has already demonstrated efficacy in HIV negative individuals with enlargement of the masseter muscle. Botulinum toxin has also been used safely in the salivary glands in individuals with excessive drooling resulting from neurological disease. In a trial HIV+ patient, the investigators have already demonstrated the efficacy of using botulinum toxin A in the treatment of posterior cheek enlargement, resulting from both parotid and masseter muscle enlargement. The investigators anticipate this study will increase our understanding of posterior cheek enlargement in HIV and lead to the development of a novel treatment for this important complication.

The investigators hypothesize that posterior cheek enlargement in HIV+ patients will in some cases result from both masseter muscle hypertrophy as well as parotid gland enlargement. The investigators also hypothesize that the treatment of posterior cheek enlargement with botulinum toxin A will result in a more aesthetically appealing lower facial contour in HIV+ patients. This has already been demonstrated in a trial HIV+ patient, in which there was a dramatic change in the volume of the masseter muscle and parotid gland 12 weeks after treatment with botulinum toxin A.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE

Altered contour of the lower face is a frequent complication of HIV and can lead to significant cosmetic disfigurement and social stigmatization. However, posterior cheek enlargement in HIV is poorly characterized. The parotid and masseter overlie the mandibular ramus, thus both contributing to the lower facial contour. Parotid hypertrophy is a recognized and common complication of HIV. It is presently unknown whether masseter muscle hypertrophy also contributes to this cosmetic deformity. The investigators will conduct a prospective pilot study in HIV+ patients to determine whether masseter muscle hypertrophy and parotid gland enlargement contribute to a bulky and widened lower facial contour, or whether the aesthetic appearance is due primarily to apparent muscle enlargement attributable to facial lipoatrophy.

Development of novel treatments to address these HIV-associated cosmetic changes is increasingly important as the burden of this disease expands globally. There have been limited advances in salivary gland surgery in recent years. The benign nature of parotid gland hypertrophy requires the surgeon to preserve key anatomical structures as an important marker of outcome. As such, parotidectomy is a controversial procedure. Treatments for masseter hypertrophy include surgical reduction of the masseter muscle and resection of the mandibular angle to create a narrower facial width. These surgical treatments can involve significant complications such as facial nerve injury, infection, scarring, bleeding, swelling and trismus. This highlights the need to develop more treatments for posterior cheek enlargement. Botulinum toxin is a highly efficacious and cost-effective, nonsurgical option for reducing the width and improving the shape of the lower face and jawline. Botulinum toxin for masseter hypertrophy and parotid enlargement in HIV negative individuals and sialorrhea in neurological disease is a safe and effective treatment for these conditions. However, there are no studies published to date on the use of botulinum toxin in the setting of HIV. Furthermore, the investigators have already demonstrated the efficacy of using botulinum toxin A in the treatment of posterior cheek enlargement in a trial HIV+ patient with both parotid enlargement and masseter hypertrophy. This patient had a dramatic response clinically and demonstrated a 19.0% and 19.4% mean reduction in the volume of the parotid gland and masseter muscle, respectively, 12 weeks after injection of botulinum toxin A. He experienced no adverse effects from the injections.

The investigators will use clinical, photographic and radiological evaluations to determine the efficacy and durability of botulinum toxin A for altered lower facial contour in HIV+ patients. The investigators anticipate that, at a minimum, this study will improve our understanding of posterior cheek enlargement seen in some HIV+ patients. The results of this study may translate into a novel and evidence-based use of botulinum toxin for management of altered lower facial contour in HIV+ patients. This could potentially improve the psychosocial wellbeing in patients afflicted with this devastating disease.

STUDY PROTOCOL

This will be an initial pilot study with 5 participants. Participants with posterior cheek enlargement will have photographs taken and a baseline CT scan of the head performed. Botulinum toxin A will be injected by identifying the inferior border of the zygomatic arch and mandibular ramus as well as the anterior and posterior demarcation of the posterior cheek enlargement. Injections will be performed percutaneously by palpation. A total of 10 U will be injected into 5 evenly spaced points of the posterior cheek enlargement to give a total dose of 50 U per side.

Participants will be evaluated clinically at 4, 8 and 12 weeks after injection, with photographs, and by a questionnaire assessing patient satisfaction and side effects. A CT scan of the head will be performed 12 weeks after injection of botulinum toxin A. Long-term efficacy of botulinum toxin A will then be evaluated at 6 and 12 months post injection clinically, with photographs and a questionnaire assessing patient satisfaction and side effects.

The primary outcome will be the change in volume of the masseter muscle and parotid gland 12 weeks after treatment with botulinum toxin A. The mean change and standard deviation will be determined. A secondary outcome will be the relative contributions of masseter hypertrophy and parotid enlargement to posterior cheek enlargement in HIV+ patients. The pre-treatment volume of the masseter muscle and parotid gland determined in our HIV+ participants will be compared to those of normal controls published in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 and older
2. Are HIV positive
3. Have facial lipoatrophy and a clinically widened lower facial contour

Exclusion Criteria:

1. Have had previous facial injection of any other products
2. Have an active infection on the face
3. Are receiving active treatment with interferon or systemic corticosteroids
4. Are pregnant or breast-feeding
5. Have known preexisting renal disease
6. Have poorly controlled diabetes mellitus

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Carruthers, MD, Principal Investigator — University of British Columbia
Locations (1):
- Carruthers Dermatology Center, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin A
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HIV Posterior Cheek Enlargement Group: Patients with HIV posterior cheek enlargement treated with botulinum toxin A
Arm/Group | HIV Posterior Cheek Enlargement Group
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
parotid gland volumes [Number; unit: participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Volume of the Masseter Muscle From Baseline to 12 Weeks After Treatment With Botulinum Toxin A
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: percentage reduction in masseter volume
Arm/Group | HIV Posterior Cheek Enlargement Group
Number analyzed (Participants) | 5
percentage reduction in masseter volume | 21.4 [10 to 27.4]

2. Primary Outcome: Percentage Change in Volume of the Parotid Gland From Baseline to 12 Weeks After Treatment With Botulinum Toxin A
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: percentage reduction in parotid volume
Arm/Group | HIV Posterior Cheek Enlargement Group
Number analyzed (Participants) | 5
percentage reduction in parotid volume | 11.2 [6.4 to 14.6]

ADVERSE EVENTS:
Groups:
- HIV Posterior Cheek Enlargement Group: Injected with botulinum toxin A
Arm/Group | HIV Posterior Cheek Enlargement Group
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV Posterior Cheek Enlargement Group (N=5)
decrease in bite force (Musculoskeletal and connective tissue disorders) | 2
change in facial expression (Skin and subcutaneous tissue disorders) | 1
dysgeusia (Gastrointestinal disorders) | 1
sunken cheeks (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This was a pilot study with only 5 participants. This study can only serve as a guide for larger studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No